CLINICAL TRIAL: NCT05616325
Title: Long-term Follow-up of Ovarian Function and Fertility in Young Lymphoma Patients Treated by Chemotherapy
Brief Title: Long-term Ovarian Fertility in Patients Treated for Lymphoma.
Acronym: FERTILymph
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Lille (Other)
Collaborators: Agence Régionale de Santé Hauts de France (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2022_0072; 2022-A01753-40 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2022-11-07; First posted 2022-11-15 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Lymphoma, Follicular
Keywords: Ovarian reserve; chemotherapy, antimüllerian hormone, lymphoma, fertility, follicle; antimüllerian hormone, lymphoma, fertility, follicle; lymphoma; follicle
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an observational, single-center, longitudinal cohort study. In order to evaluate the gonadotoxicity of chemotherapy, an AMH monitoring was initiated in 2006 in our fertility observatory in young patients with lymphoma before, during and after chemotherapy. This study is part of the project "She will get better and then want a child" and is supported by the ARS hauts de France (n° DOS/SDES/AR/FIR/2019/282). Our first study published in 2010 shows that AMH decreases sharply during chemotherapy, regardless of the chemotherapy protocol. At the end of chemotherapy, AMH recovery profiles differ according to the protocol received. This follow-up is therefore essential in order to adapt our practices and our preservation strategies, particularly to the type of chemotherapy. Patients are primarily concerned about their chances of subsequent pregnancy, and there is little evidence in the literature about the impact of chemotherapy on ovarian reserve and long-term fertility.

The fisrt objective of our study is to evaluate, at distance from chemotherapy, the evolution of ovarian function in patients treated for lymphoma by evaluating follicular reserve parameters (AMH and antral follicle count) at 5 and 10 years after the end of chemotherapy compared with the initial workup performed before chemotherapy and the workup performed at 12 months after the end of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a history of lymphoma treated with chemotherapy
* followed in the fertility observatory of the Jeanne de Flandre Hospital at the University Hospital of Lille (project "she will heal and then want a child"), who are at least at 5 years since the end of chemotherapy
* Patients having been informed and having given their written consent to participate in the study.
* Beneficiary of a social security system.

Exclusion Criteria:

* Patient not followed in the fertility observatory.
* Inability of the patient to undergo the medical follow-up of the trial for geographical, social or psychological reasons.
* Patient opposed to her participation in the study.
* Patient under guardianship or curatorship.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — women of childbearing age
Study Population: lymphoma patients treated with chemotherapy included in the fertility observatory
Sampling Method: Probability Sample
Enrollment: 270 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2029-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Follicular reserve parameters (AMH and antral follicle count) | at the end of chemotherapy
  Follicular reserve parameters (AMH and antral follicle count) at 5 and 10 years after the end of chemotherapy compared with the initial workup performed before chemotherapy and the workup performed at 12 months after the end of chemotherapy

SECONDARY OUTCOMES:
Cumulative incidence of pregnancy at 5 years and 10 years from the end of treatment defined by the achievement of at least one spontaneous or induced pregnancy. | at 5 and 10 years after the end of chemotherapy.
Pregnancy rate obtained by ART (with or without gamete reuse) | at 5 and 10 years after the end of chemotherapy.
  defined by the ratio between the number of clinical pregnancies and the number of ART attempts performed (with or without gamete reuse or frozen ovarian tissue).
Rate of miscarriages, ectopic pregnancies, and live births (single, multiple) | at 5 and 10 years after the end of chemotherapy.
  defined by the ratio of the number of miscarriages, ectopic pregnancies, and live births to the number of pregnancies obtained by ART (with or without reuse of gametes or frozen ovarian tissue).
Scores on the Reproductive Concerns (RCACS) | at 5 and 10 years after the end of chemotherapy.
Scores Mood (PHQ) | at 5 and 10 years after the end of chemotherapy.
Quality of Life (FACT-G7) | at 5 and 10 years after the end of chemotherapy.
Life Satisfaction (SWLS) scales | at 5 and 10 years after the end of chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Christine DECANTER, MD,PhD, Principal Investigator — University Hospital, Lille